CLINICAL TRIAL: NCT06237101
Title: Influence of Variable Plasma Concentrations of Remifentanil on Burst Suppression (BS) Event Rate in Electroencephalographic (EEG) Recordings of Human Subjects Undergoing Total Intravenous General Anesthesia (TIVA) Under Propofol
Brief Title: Remifentanil Effect on Burst Suppression Ratio
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: OAIC: 1345/23
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Anesthesia, Intravenous; Electroencephalography; Burst Suppression
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High dose (Experimental): Propofol concentration which generate burst suppression at high dose of remifentanil
  Interventions: Drug: High dose of remifentanil
- Medium dose (Active Comparator): Propofol concentration which generate burst suppression at medium dose of remifentanil
  Interventions: Drug: Medium dose of remifentanil

INTERVENTIONS:
Drug: High dose of remifentanil — The dose of remifentanil will be changed to determine the concentration of propofol at which burst suppressions are generated
  Arms: High dose
Drug: Medium dose of remifentanil — The dose of remifentanil will be changed to determine the concentration of propofol at which burst suppressions are generated
  Arms: Medium dose

SUMMARY:
The goal of this clinical trial is to determine whether remifentanil has a facilitating effect on the generation of burst suppression by propofol in adult patients (18-60 years) candidates for elective surgery who require remifentanil and American Society of Anesthesiology (ASA) classification I or II. The main question it aims to answer are:

• To determine whether remifentanil has a facilitating effect on the generation of burst suppression by propofol.

Participants will undergo general anesthesia with remifentanil and propofol sequentially. After loss of consciousness, remifentanil will be adjusted to a medium or high concentration randomly and it will be determined at what concentration of propofol the burst suppressions are generated.

Then, the concentrations of propofol that generate burst suppression associated with either a medium or high concentration of remifentanil will be compared.

DETAILED DESCRIPTION:
Subjects will enter the ward, after which an 18 G intravenous cannula will be installed and will be monitored under the routinely applied ASA standard. Frontal EEG activity will be recorded using an anesthetic depth monitor and a baseline EEG will be recorded for 120 seconds with eyes closed. Subjects will then be preoxygenated. Once the oxygen concentration at the end of expiration reaches 90%, the administration of remifentanil will begin, under the Minto pharmacological model, to reach an effect site concentration of 7.5 ng/mL. Once the remifentanil concentration is reached, the infusion of propofol will begin at a rate of 15 mg/kg/h using Base Primea Orchestra, until loss of consciousness (LOC) is achieved. LOC will be defined as loss of response to verbal and tactile stimulation, which will be corroborated every 30 seconds. After this, the propofol infusion will be maintained at the concentration at which the LOC occurred, based on Marsh's pharmacological model, and rocuronium 0.6 mg/kg will be administered to facilitate orotracheal intubation.

Once the patient has been intubated, the remifentanil will be lowered to a concentration of 4 ng/mL and the surgery will continue. After 5 min after the LOC occurred, according to randomization, the concentration of remifentanil will remain at 4 ng/mL or increase to 7.5 ng/mL, and 10 min after the LOC occurred the propofol infusion rate will be changed to 15 mg/kg/h for 10 min. After this, the propofol concentration at which the LOC occurred will be returned and remifentanil will be maintained at 4 ng/mL. After 5 min after completing the previous step, remifentanil will be increased to 7.5 ng/mL or maintained at 4 ng/mL in the opposite way to what happened previously. After 10 min after completing the previous step, propofol will be dosed again at a fixed rate of 15 mg/kg/h for 10 min. Finally, after this time has elapsed, the concentration of propofol at which the LOC occurred will be returned and the remifentanil will be dosed according to the surgical requirements. Throughout the protocol, hemodynamics will be maintained with the usual management of drugs such as ephedrine in boluses or norepinephrine in continuous infusion.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology I or II
* Elective surgery of low or intermediate risk

Exclusion Criteria:

* Neurological disease
* Psychiatric disease
* Use of psychoactive drugs or opioids
* Altered basal state of consciousness
* Allergy to propofol
* Body mass index > 35 kg/m2
* Pre-existing renal, cardiac and/or hepatic dysfunction
* Patient's refusal to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Propofol estimated concentration by Marsh pharmacological model, which generates burst suppression | During 10 minutes when propofol dosification is increased to 15 mg/kg/h
  [mcg/mL]

SECONDARY OUTCOMES:
Propofol estimated concentration by Marsh pharmacological model, which generates loss of consciousness | Minutes, during anesthesia induction is performed
  [mcg/mL]
Mean arterial pressure during burst suppression | During 10 minutes when propofol dosification is increased to 15 mg/kg/h
  mmHg
Total ephedrine dose | During all protocol, 40 min
  mg
Maximal dose of norepinephrine | During all protocol, 40 min
  mcg/kg/min
Bispectral index at burst suppression | During 10 minutes when propofol dosification is increased to 15 mg/kg/h
  (0-100), 0 indicates a flat electroencephalogram and 100 indicates to be awake.

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - Centro de Investigación Cínica Avanzada (CICA), Hospital Clinico de la Universidad de Chile, Santiago, RM
  - Hospital Clinico de la Universidad de Chile, Santiago, RM